CLINICAL TRIAL: NCT02053480
Title: Pyruvate Kinase Deficiency (PKD) Natural History Study
Brief Title: Pyruvate Kinase Deficiency Natural History Study
Acronym: PKD NHS
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Rachael Grace, Principal Investigator, PKD Natural History Study, Boston Children's Hospital
Other Study IDs: P00010515
Record Dates: First submitted 2014-01-28; First posted 2014-02-03 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Pyruvate Kinase Deficiency; Congenital Non-Spherocytic Hemolytic Anemia
Keywords: pyruvate kinase deficiency; hemolytic anemia; anemia; enzymopathy; jaundice; splenectomy; health-related quality of life; Hematologic diseases
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic; Anemia; Jaundice; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pyruvate Kinase Deficiency: Patients of all ages with Pyruvate Kinase Deficiency

SUMMARY:
The purpose of this study is to describe the range and incidence of symptoms, treatments, and complications related to pyruvate kinase deficiency (PKD). Eligible patients are those of all ages with known PKD or with a hemolytic anemia and a family member with PKD. The study will collect retrospective medical history, routine clinical care data, and quality of life measures at baseline and annually for patients with PKD.

DETAILED DESCRIPTION:
The purpose of the Pyruvate Kinase Deficiency (PKD) Natural History Study is to describe the natural history of PKD and the range and incidence of symptoms, treatments, and complications related to PKD. The study will collect retrospective medical history and routine clinical care data at baseline and annually for patients with PKD. Patients without a genetic diagnosis will have a blood sample drawn for genetic diagnostic confirmation for research purposes. Understanding the clinical variation among participants with PKD, and assessing treatments specific to PKD and their outcomes will accelerate improvement in the care of patients with PKD. Understanding the natural history of PKD may be useful in the design of future interventional studies. Detailed genotypic and phenotypic characterization of the cohort will allow for continued in depth characterization of PKD. Finally, the PKD Natural History Study will identify interested participants for future PKD studies.

Primary Objectives:

1. To estimate the transfusion burden in splenectomized and non-splenectomized participants with PKD.
2. To establish a patient registry as a potential source for recruitment to future research studies in PKD.

Secondary Objectives:

1. To determine if patient-reported outcomes, including quality of life and fatigue scales, are associated with age, genotype, hemoglobin nadir, and/or transfusion burden, overall and within the subgroups of splenectomized vs. non-splenectomized participants;
2. To describe changes over time in the range of hemoglobin values and markers of hemolysis within individual participants and among participants with PKD;
3. To estimate the incidence of past splenectomy and annual splenectomy rate, as treatment for PKD;
4. To estimate the prevalence and severity and describe the treatment of hepatic and cardiac iron overload and its complications in PKD (liver, cardiac, growth defects, hypogonadotropic hypogonadism, and other endocrine defects). To describe the changes in these complications that may occur over time and by age group;
5. To estimate the prevalence of co-morbidities associated with chronic hemolysis in PKD, to identify which co-morbidities are the most common, and to determine if the prevalence and/or severity of co-morbidities change over time and by age at the time of the first appearance of the co-morbidity;
6. To determine pregnancy outcomes among participants with PKD;
7. To describe genotypic and phenotypic variation among participants and explore genotype-phenotype correlation in PKD.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages with biochemically or genetically diagnosed PKD.
* Patients with a hemolytic anemia AND a family member with genetically diagnosed PKD
* The participant or the guardian of the participant is willing and able to give written informed consent and/or assent.

Exclusion Criteria:

* The participant or the guardian of the participant is unwilling or unable to give written informed consent and/or assent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Pyruvate Kinase Deficiency of all ages
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2013-12; Primary Completion 2019-12 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
transfusion burden in splenectomized and non-splenectomized participants | 12 weeks

SECONDARY OUTCOMES:
patient-reported outcomes | enrollment, annually, up to 2 years
  EuroQoL-5D-5L, Functional Assessment of Cancer Therapy-Anemia (FACT-An), Pediatric Quality of Life Inventory 4.0 (pedsQL 4.0), Pediatric Functional Assessment of Chronic Illness-Fatigue (pedsFACIT-F), Patient Reported Outcomes Measurement Information System Fatigue (PROMIS Fatigue)
changes over time in hemoglobin and markers of hemolysis | enrollment, annually, up to 2 years
prevalence and severity of iron overload | enrollment, annually, up to 2 years

CONTACTS AND LOCATIONS:
Locations (30):
- United States (19):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - DDC Clinic for Special Needs Children, Middlefield, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Central Pennsylvania Clinic, Strasburg, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont College of Medicine & University of Vermont Medical Center, Burlington, Vermont
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Fakultni Nemocnice Olomouc, Olomouc, Czechia
- Germany (5):
  - Charite Berlin, Berlin
  - University of Freiburg, Freiburg im Breisgau
  - UniversitätsKlinikum Heidelberg, Zentrum für Kinder- und Jugendmedizin Klinik Kinderheilkunde III, Heidelberg
  - Klinikum Kassel, Kassel
  - Klinikum der Universität München, Center for Pediatric Hematology/Hemostaseology, Munich
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grace RF, Bianchi P, van Beers EJ, Eber SW, Glader B, Yaish HM, Despotovic JM, Rothman JA, Sharma M, McNaull MM, Fermo E, Lezon-Geyda K, Morton DH, Neufeld EJ, Chonat S, Kollmar N, Knoll CM, Kuo K, Kwiatkowski JL, Pospisilova D, Pastore YD, Thompson AA, Newburger PE, Ravindranath Y, Wang WC, Wlodarski MW, Wang H, Holzhauer S, Breakey VR, Kunz J, Sheth S, Rose MJ, Bradeen HA, Neu N, Guo D, Al-Sayegh H, London WB, Gallagher PG, Zanella A, Barcellini W. Clinical spectrum of pyruvate kinase deficiency: data from the Pyruvate Kinase Deficiency Natural History Study. Blood. 2018 May 17;131(20):2183-2192. doi: 10.1182/blood-2017-10-810796. Epub 2018 Mar 16. PMID 29549173
- [Background] van Beers EJ, van Straaten S, Morton DH, Barcellini W, Eber SW, Glader B, Yaish HM, Chonat S, Kwiatkowski JL, Rothman JA, Sharma M, Neufeld EJ, Sheth S, Despotovic JM, Kollmar N, Pospisilova D, Knoll CM, Kuo K, Pastore YD, Thompson AA, Newburger PE, Ravindranath Y, Wang WC, Wlodarski MW, Wang H, Holzhauer S, Breakey VR, Verhovsek M, Kunz J, McNaull MA, Rose MJ, Bradeen HA, Addonizio K, Li A, Al-Sayegh H, London WB, Grace RF. Prevalence and management of iron overload in pyruvate kinase deficiency: report from the Pyruvate Kinase Deficiency Natural History Study. Haematologica. 2019 Feb;104(2):e51-e53. doi: 10.3324/haematol.2018.196295. Epub 2018 Sep 13. No abstract available. PMID 30213831
- [Background] Bianchi P, Fermo E, Lezon-Geyda K, van Beers EJ, Morton HD, Barcellini W, Glader B, Chonat S, Ravindranath Y, Newburger PE, Kollmar N, Despotovic JM, Verhovsek M, Sharma M, Kwiatkowski JL, Kuo KHM, Wlodarski MW, Yaish HM, Holzhauer S, Wang H, Kunz J, Addonizio K, Al-Sayegh H, London WB, Andres O, van Wijk R, Gallagher PG, Grace RFF. Genotype-phenotype correlation and molecular heterogeneity in pyruvate kinase deficiency. Am J Hematol. 2020 May;95(5):472-482. doi: 10.1002/ajh.25753. Epub 2020 Mar 6. PMID 32043619
- [Derived] Al-Samkari H, van Beers EJ, Morton DH, Eber SW, Chonat S, Kuo KHM, Kollmar N, Wang H, Breakey VR, Sheth S, Sharma M, Forbes PW, Klaassen RJ, Grace RF. Health-related quality of life and fatigue in children and adults with pyruvate kinase deficiency. Blood Adv. 2022 Mar 22;6(6):1844-1853. doi: 10.1182/bloodadvances.2021004675. PMID 34470054